CLINICAL TRIAL: NCT02475499
Title: The Use of Incretin-based Drugs and the Risk of Pancreatic Cancer in Patients With Type 2 Diabetes
Brief Title: Incretin-based Drugs and Pancreatic Cancer
Status: Completed | Type: Observational
Sponsor: Canadian Network for Observational Drug Effect Studies, CNODES (Other)
Collaborators: Drug Safety and Effectiveness Network, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: Q13-06A
Record Dates: First submitted 2015-06-16; First posted 2015-06-18 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Incretins; Antidiabetic agents; Pancreatic Cancer
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Pancreatic Neoplasms | interventions — Dipeptidyl-Peptidase IV Inhibitors; Sitagliptin Phosphate; Vildagliptin; saxagliptin; Glucagon-Like Peptide-1 Receptor Agonists; Exenatide; Liraglutide; Sulfonylurea Compounds; Hypoglycemic Agents; Glyburide; Chlorpropamide; Tolbutamide; glibornuride; Tolazamide; Carbutamide; Glipizide; gliquidone; Gliclazide; metahexamide; glisoxepide; glimepiride; Acetohexamide; glymidine; Biguanides; Phenformin; Metformin; Buformin; Thiazolidinediones; Troglitazone; Rosiglitazone; Pioglitazone; Glycoside Hydrolase Inhibitors; Acarbose; miglitol; voglibose; meglitinide; repaglinide; Nateglinide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Treated with incretins: Ever-use of incretin-based drugs ((DPP-4 inhibitors [sitagliptin, vildagliptin, and saxagliptin] or GLP-1 analogs [exenatide, liraglutide]) between (and including) base cohort entry and the index day - 365 days.
  Interventions: Drug: DPP-4 inhibitors; Drug: GLP-1 analogs
- Treated with sulfonylureas: Ever-use of sulfonylureas between (and including) base cohort entry and the index day - 365 days, and never-use of incretin-based drugs.
  Interventions: Drug: Sulfonylureas
- Treated with other antidiabetic agents: Ever-use of other antidiabetic agents (biguanides, thiazolidinediones, alpha-glucosidase inhibitors, meglitinides) between (and including) base cohort entry and the index day - 365 days, with never-use of incretin-based drugs and never use of sulfonylureas.
  Interventions: Drug: Biguanides; Drug: Thiazolidinediones; Drug: Alpha-glucosidase inhibitors; Drug: Meglitinides

INTERVENTIONS:
Drug: DPP-4 inhibitors — Ever-use of DPP-4 inhibitors (ATC A10BH, A10BD07-A10BD13) will be defined as a prescription occurring between (and including) base cohort entry and the index day - 365 days.
  Other Names: incretin-based drugs; sitagliptin; vildagliptin; saxagliptin
  Groups: Treated with incretins
Drug: GLP-1 analogs — Ever-use of GLP-1 analogs (ATC A10BX04, A10BX07) will be defined as a prescription occurring between (and including) base cohort entry and the index day - 365 days.
  Other Names: incretin-based drugs; exenatide; liraglutide
  Groups: Treated with incretins
Drug: Sulfonylureas — Ever-use of sulfonylureas (ATC A10BB or A10BC) will be defined as a prescription occurring between (and including) base cohort entry and the index day - 365 days.
  Other Names: oral hypoglycemic agent; glibenclamide; chlorpropamide; tolbutamide; glibornuride; tolazamide; carbutamide; glipizide; gliquidone; gliclazide; metahexamide; glisoxepide; glimepiride; acetohexamide; glymidine
  Groups: Treated with sulfonylureas
Drug: Biguanides — Ever-use of biguanides (ATC A10BA) will be defined as a prescription occurring between (and including) base cohort entry and the index day - 365 days.
  Other Names: oral hypoglycemic agent; phenformin; metformin; buformin
  Groups: Treated with other antidiabetic agents
Drug: Thiazolidinediones — Ever-use of thiazolidinediones (ATC A10BG) will be defined as a prescription occurring between (and including) base cohort entry and the index day - 365 days.
  Other Names: oral hypoglycemic agent; troglitazone; rosiglitazone; pioglitazone
  Groups: Treated with other antidiabetic agents
Drug: Alpha-glucosidase inhibitors — Ever-use of alpha-glucosidase inhibitors (ATC A10BF) will be defined as a prescription occurring between (and including) base cohort entry and the index day - 365 days.
  Other Names: oral hypoglycemic agent; acarbose; miglitol; voglibose
  Groups: Treated with other antidiabetic agents
Drug: Meglitinides — Ever-use of meglitinides (ATC A10BX02, A10BX03) will be defined as a prescription occurring between (and including) base cohort entry and the index day - 365 days.
  Other Names: oral hypoglycemic agent; repaglinide; nateglinide
  Groups: Treated with other antidiabetic agents

SUMMARY:
The purpose of this study is to determine whether incretin-based drugs (used to treat type 2 diabetes) taken either alone in or combination with other anti-diabetic drugs are associated with an increased risk of pancreatic cancer (PC) compared to sulfonylureas.

The investigators will carry out separate population based cohort studies using administrative health databases in five jurisdictions in Canada, the US, and the UK. Cohorts will be defined by the initiation of a new anti-diabetic drug when incretin-based drugs entered the market, with follow-up until hospitalization for PC. The results from the separate sites will be combined to provide an overall assessment of the risk of PC in users of incretin-based drugs and by class of incretin-based drugs.

DETAILED DESCRIPTION:
The study objective is to determine whether the use of incretin-based drugs, compared with the use of sulfonylureas, is associated with an increased risk of pancreatic cancer (PC) in routine clinical practice. The investigators will use a common-protocol approach to conduct retrospective cohort studies using administrative health care data from five jurisdictions (the Canadian provinces of Alberta, Manitoba, and Ontario, as well as United States (US) MarketScan, and the United Kingdom (UK) Clinical Practice Research Datalink [CPRD]). Briefly, the Canadian databases include population-level data on physician billing, diagnoses and procedures from hospital discharge abstracts, and dispensations for prescription drugs. Ontario data will be restricted to patients aged 65 years and older as prescription data are not available for younger patients. The CPRD is a clinical database that is representative of the UK population and contains the records for patients seen at over 680 general practitioner practices in the UK; these data will be linked to the Hospital Episode Statistics (HES) database, which contains in-hospital diagnosis and procedure data. US MarketScan includes individuals and their dependents covered by large U.S. employer health insurance plans, and government and public organizations.

Study population

In each jurisdiction, the investigators will assemble a base cohort that includes all patients with a first-ever prescription for a non-insulin anti-diabetic drug, including biguanides, sulfonylureas, thiazolidinediones, DPP-4 inhibitors, GLP-1 analogs, alpha-glucosidase inhibitors, meglitinides, or combinations of these drugs from the earliest availability of data at each site to the last date of availability of data. The date of prescription (for the CPRD) or dispensation (for all other sites) of the first-ever non-insulin anti-diabetic drug will define the date of base cohort entry. From this base cohort, a study cohort will be created including all patients who initiated a new anti-diabetic drug class during the year in which incretin-based drugs entered the market in each jurisdiction or any time thereafter. These new users consist of both those who are newly-treated for diabetes, as well as those who switch to or add on a new anti-diabetic drug class not included as part of their previous treatment history. The date of study cohort entry is defined by the prescription date of the newly-prescribed drug class. Patients in the study cohort will be followed from the date of study cohort entry + 365 days until an event (defined below) or censoring due to death, departure from the database, loss of continuous health plan or drug plan enrolment, entry into a long-term care facility, or the end of the study period (June 30, 2014 or the last date of data availability at that site), whichever occurs first.

Case-control selection

The cohort defined above will be analyzed using a nested case-control analysis, where cases are defined as a hospitalization for PC. Risk set sampling will be used to randomly select up to 20 controls for each case, matched on sex, age (± 365 days), date of study cohort entry (± 180 days), duration of treated diabetes (± 90 days), and duration of follow-up in days.

Exposure assessment

Ever-use of an anti-diabetic drug will be defined as any prescription for an anti-diabetic agent between base cohort entry and the index day -365 days. This 365-day lag period will be applied to account for disease latency and potential protopathic bias by only considering prescriptions received from (and including) the Base Cohort Entry Date until (and including) the date one year prior to the Index day. Ever-use of exposure will be classified hierarchically based on the following three mutually-exclusive categories: 1) incretin-based drugs; 2) sulfonylureas; 3) other antidiabetic agents. Sulfonylureas will serve as the primary reference category as incretin-based drugs are second- to third-line therapy and thus used at a comparable point in the disease management.

Statistical analyses

Conditional logistic regression will be used to estimate odds ratios (ORs) and corresponding 95% confidence intervals (CIs) of the association of hospitalization for PC, comparing ever-use of incretin-based drugs to ever-use of sulfonylureas. This is considered the primary analysis. Secondary analyses will include sub-classifying ever-users of incretin-based drugs by type (i.e., DPP-4 inhibitor vs GLP-1 analog), cumulative duration of ever-use (≤ 365 days, 366-729 days, and ≥730 days), and time since initiation of treatment among ever-users. In addition, four sensitivity analyses will be conducted, all defined a priori, to assess the robustness of the results. Finally, all site-specific estimates will be meta-analyzed using random-effects models with inverse variance weighting, with fixed-effects analyses conducted as sensitivity analyses. The amount of between-site heterogeneity will be estimated using the I square statistic.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a first-ever prescription for a non-insulin anti-diabetic drug, including biguanides, sulfonylureas, thiazolidinediones, DPP-4 inhibitors, GLP-1 analogs, alpha-glucosidase inhibitors, meglitinides or combinations of these drugs from the earliest availability of data at each site to the last date of availability of data.
* Patients with at least 1 year of history in the database.
* Patients at least 18 years of age.

Exclusion Criteria:

* Patients who died or left the cohort before the year the first incretin-based drug entered the market.
* Patients who never added-on or switched to a new anti-diabetic drug after incretin-based drugs entered the market up until June 30, 2014.
* Patients with a previous diagnosis of pancreatic cancer, those who underwent pancreatectomy or were diagnosed with congenital defects of the pancreas at any time prior to study cohort entry.
* Patients with less than 365 days of follow-up after study cohort entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In each jurisdiction, a base cohort will be assembled including all patients with a first-ever prescription for a non-insulin anti-diabetic drug. Base cohort entry is defined as the date of prescription or dispensation of the first-ever non-insulin anti-diabetic drug. From this base cohort, a study cohort will be formed consisting of all patients who initiated a new anti-diabetic drug class during the year in which incretin-based drugs entered the market in each jurisdiction or any time thereafter. Study cohort entry is defined by the prescription date of the newly-prescribed drug class.
Sampling Method: Probability Sample
Enrollment: 886172 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Incident pancreatic cancer | Patients were followed from the date of study cohort entry until hospitalization for incident pancreatic cancer, censoring, or for up to 79 months.
  Incident cases of pancreatic cancer recorded in a hospital database with the following ICD codes:
  ICD-9:157.0-157.9
  ICD-10:C25.x

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Ernst, MD, MSc, Principal Investigator — Lady Davis Institute for Medical Research, Jewish General Hospital - McGill University
Locations (1):
- Lady Davis Institute for Medical Research, Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Result] Azoulay L, Filion KB, Platt RW, Dahl M, Dormuth CR, Clemens KK, Durand M, Juurlink DN, Targownik LE, Turin TC, Paterson JM, Ernst P; Canadian Network for Observational Drug Effect Studies Investigators. Incretin based drugs and the risk of pancreatic cancer: international multicentre cohort study. BMJ. 2016 Feb 17;352:i581. doi: 10.1136/bmj.i581. PMID 26888382
- See also: This organization's website describing general functions, other CNODES projects, and investigator profiles. — http://www.cnodes.ca